CLINICAL TRIAL: NCT03231033
Title: First in Human Study of Pioglitazone Therapy of Autoimmune Pulmonary Alveolar Proteinosis
Brief Title: Pioglitazone Therapy of Autoimmune Pulmonary Alveolar Proteinosis Autoimmune Pulmonary Alveolar Proteinosis
Acronym: PioPAP
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: TPSC-114
Record Dates: First submitted 2017-06-19; First posted 2017-07-27 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2019-01

CONDITIONS: Autoimmune Pulmonary Alveolar Proteinosis
MeSH Terms: conditions — Pulmonary Alveolar Proteinosis, Acquired | interventions — Pioglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pioglitazone (Experimental): Oral administration of Actos at 15 mg/day for 12 weeks, 30 mg/day for 12 weeks, and 45 mg/day for 12 weeks
  Interventions: Drug: Pioglitazone

INTERVENTIONS:
Drug: Pioglitazone — Participants will receive three doses of Pioglitazone, 15 mg/day for 12 weeks, 30 mg/day for 12 weeks, and 45 mg/day for 12 weeks
  Other Names: Actos

SUMMARY:
Pulmonary alveolar proteinosis (PAP) is a syndrome of surfactant accumulation, respiratory failure, and innate immune deficiency for which therapy remains limited to whole lung lavage (WLL), an invasive physical procedure to remove surfactant unavailable at most medical centers. While PAP occurs in multiple diseases affecting men, women, and children of all ages and ethnic origins, in 85% of patients, it occurs as an idiopathic disease associated with neutralizing GM-CSF autoantibodies. Basic science and translational research has shown that idiopathic PAP is an autoimmune disease in which disruption of GM-CSF signaling impairs the ability of alveolar macrophages to clear surfactant and perform host defense functions.

Recently, it has been shown that cholesterol toxicity drives pathogenesis in alveolar macrophages from GM-CSF deficient (Csf2-/-) mice and patients with autoimmune PAP. Loss of GM-CSF signaling reduces PU.1/CEBP-mediated expression of PPARγ and its downstream target ABCG1 (a cholesterol exporter important in macrophages). The cell responds by esterifying and storing cholesterol in vesicles to reduce toxicity. Eventually, vesicles fill the cell, impair intracellular transport and reduce uptake and clearance of surfactant from the lung surface resulting in disease manifestations. Recent data indicates that pioglitazone, a PPARγ agonist currently approved by the FDA for human use, increases cholesterol/surfactant clearance by alveolar macrophages from autoimmune PAP patients and Csf2-/- mice. Importantly, pioglitazone significantly reduced the severity of PAP lung disease in Csf2-/- mice after several months of therapy. Together, these observations suggest pioglitazone could be 'repurposed' as pharmacologic therapy for PAP.

DETAILED DESCRIPTION:
PAP is a rare syndrome of surfactant accumulation and resulting hypoxemic respiratory failure that occurs in multiple diseases that can be classified on the basis of pathogenesis into three groups: primary PAP (caused by disruption of GM-CSF signaling - autoimmune PAP, hereditary PAP), secondary PAP (caused by reduction in alveolar macrophage numbers and/or functions), and metabolic disorders of surfactant production-related PAP (caused by mutations in genes required for normal surfactant production). Blood tests are capable of identifying the PAP-causing disease in about 95% of patients.

Research has demonstrated that aPAP is caused by a high level of GM-CSF autoantibodies, which block GM-CSF signaling. Normally, alveolar macrophages clear (remove) about half of the used surfactant from air sacs (alveoli) in the lungs. Without GM-CSF, alveolar macrophages have a reduced ability to clear surfactant, which builds up in the alveoli and the blocks delivery of oxygen into the blood, resulting in a low blood oxygen level and a reduced oxygen delivery to tissues of the body. This macrophage defect is thought to occur because loss of GM-CSF stimulation causes reduced activity of PPAR-gamma, a molecule present within alveolar macrophages that they require to simulate the ability to clear surfactant: the reduction in PPAR-gamma activity cause a functional impairment of surfactant clearance by alveolar macrophages.

Currently, no pharmacologic agent has been FDA-approved as therapy aPAP: it is currently treated by whole lung lavage, a procedure requiring general anesthesia and a breathing machine the lungs are individually filled with saline and drained repeatedly to physically remove the excess surfactant. Recent research has shown that pioglitazone, a drug that activates PPAR-gamma, is able to increase the ability of cultured macrophages to clear surfactant in the laboratory and that oral administration is able to reduce lung disease severity and be well-tolerated in a mouse model of aPAP. Currently, pioglitazone is approved by the FDA for treatment of increased blood sugar in patients with diabetes.

This study is a pilot phase I/II human clinical trial of oral pioglitazone as therapy for autoimmune PAP. The target population is adults with aPAP who have measurable, clinically significant disease satisfying all of the inclusion and exclusion criteria. The study design will involve recruitment, screening, and enrollment of participants into a phase I, open-label, dose-escalating, single site study. Oral pioglitazone will be administered to autoimmune PAP patients with a personalized dose escalation plan beginning at 15 mg per day, advancing to 30 mg per day and then 45 mg per day, if tolerated, in 12 week increments. Adverse events (AEs), serious AEs (SAEs), and pharmacodynamics (PD) parameters will be evaluated. The experimental approach will evaluate 1) safety of oral pioglitazone by documenting occurrence of treatment-emergent AEs and SAEs, 2) physiological effects of oral pioglitazone by measuring changes in the physiological, clinical, and quality of life parameters and 3) biochemical effects of pioglitazone on the transcriptome, phenotype, and function of mononuclear phagocytes (alveolar macrophages and monocytes) from autoimmune PAP patients. Anticipated results will determine the safety, efficacy, and biochemical effects of oral pioglitazone in patients with autoimmune PAP. These results will impact the field by 1) monitoring safety of oral pioglitazone in autoimmune PAP patients, 2) translating existing preclinical data in humans, and 3) demonstrating the results of pioglitazone in a personalized treatment plan with dose escalation in a pilot trial to evaluate the efficacy of oral pioglitazone for aPAP.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age ≥ 18 years and ≤ 80 years
* Able to understand and willing to sign a written informed consent document
* Able and willing to complete administration of study drug at home
* Able and willing to adhere to study visit schedule and study procedures
* Diagnosis of aPAP determined by:

  * History of a diagnosis of PAP with or without supporting lung histology or BAL/cytology and
  * Abnormal serum GM-CSF autoantibody test (GMAb ELISA Test) and
  * Chest CT findings compatible with a diagnosis of aPAP
* Evidence of impaired GM-CSF signaling demonstrated by an abnormal STAT5 phosphorylation index (STAT5-PI) test measured in heparinized whole blood at the time screening
* A-aDO2 ≥ 25 mm Hg

Exclusion Criteria:

* Diagnosis of any other PAP-causing disease
* aPAP complicated by:

  * Severe disease at screening/enrollment (A-aD02<55)
  * Clinically significant pulmonary fibrosis
* History of any clinically significant:

  * Other lung disease
  * Cardiovascular disease
  * Disease requiring use of systemic steroids in past year
  * History of Diabetes Mellitus
  * History of untreated osteoporosis
  * History of bladder cancer
  * Active / serious lung or systemic infection
  * Persistent or unexplained fever >101oF within 2 months of study
  * Treatment with an investigational therapeutic agent for aPAP within 3 months prior to enrollment, which includes inhaled GM-CSF
  * Abnormal clinical and/or laboratory parameters at screening
  * Women who are pregnant or plan to become pregnant
  * Concomitant or recent use of specific medicines

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2017-08-17 (Actual); Primary Completion 2019-04-02 (Actual); Study Completion 2019-04-02 (Actual)

PRIMARY OUTCOMES:
Occurrence of any treatment-emergent adverse events and serious adverse events | 1 year
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0

SECONDARY OUTCOMES:
Alveolar-arterial oxygen concentration gradient (A-aDO2) | 1 year
  Change from Baseline (Day 0) in the A-aDO2 gradient as measured at the End of Treatment
PaO2 | 1 year
  Change from Baseline (Day 0) in the PaO2 as measured at the End of Treatment
Minimum SpO2 during a standardized treadmill exercise test | 1 year
  Change from Baseline (Day 0) in the minimum SpO2 during a treadmill exercise test as measured at the End of Treatment
Time during a standardized treadmill exercise test required for SpO2 to fall below 88% (or discontinuance of testing due to dyspnea) | 1 year
  Change from Baseline (Day 0) in the time for the SpO2 to fall below 88% during the treadmill exercise test as measured at the End of Treatment
DLCO (Diffusion capacity of the lung for carbon monoxide) | 1 year
  Change from Baseline (Day 0) in the DLCO as measured at the End of Treatment
Parenchymal lung density determined by quantitative computed tomography (CT) densitometry | 1 year
  Change from Baseline (Day 0) in the parenchymal densitometry as measured at the End of Treatment
Quality of Life measured by SF-36 | 1 year
  Change from Baseline (Day 0) in the quality of life as measured at the End of Treatment
Quality of Life measured by St. George's Respiratory Questionnaire | 1 year
  Change from Baseline (Day 0) in the quality of life as measured at the End of Treatment
Shortness of breath measured by San Diego Dyspnea Score | 1 year
  Change from Baseline (Day 0) in the quality of life as measured at the End of Treatment

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Trapnell, MD, Study Director — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States